CLINICAL TRIAL: NCT02997020
Title: Ivacaftor for Acquired CFTR Dysfunction in Chronic Rhinosinusitis (EDSPD Protocol)
Status: Active, not recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Brad Woodworth, MD, Professor of Otolaryngology, University of Alabama at Birmingham
Other Study IDs: IRB-160516002; 1R01HL133006 (NIH)
Record Dates: First submitted 2016-12-14; First posted 2016-12-19 (Estimated); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: CRS

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (2):
- CRS Patients: Endoscopically-directed sinus potential difference (EDSPD) will be conducted in either the operating room or in the rhinology clinic setting to quantify CFTR activity in the sinus cavities. The potential difference will be monitored in actively inflamed areas as judged by endoscopy in comparison to an agar-filled reference butterfly electrode placed in the volar aspect of the forearm. A stable potential with the mean value of a 10-s scoring interval after perfusion of each solution will be recorded by a blinded investigator.
  Interventions: Other: EDSPD
- Control Patients: Endoscopically-directed sinus potential difference (EDSPD) will be conducted in either the operating room or in the rhinology clinic setting to quantify CFTR activity in the sinus cavities. The potential difference will be monitored in actively inflamed areas as judged by endoscopy in comparison to an agar-filled reference butterfly electrode placed in the volar aspect of the forearm. A stable potential with the mean value of a 10-s scoring interval after perfusion of each solution will be recorded by a blinded investigator.
  Interventions: Other: EDSPD

INTERVENTIONS:
Other: EDSPD — The equipment & conditions for measuring bioelectric changes across the sinus mucosa are based on the standard NPD protocol, including use of agar-filled PE90 tubing for the probing electrode and limiting perfusion solutions to Ringer, Ringer + amiloride (100 µM), chloride-free gluconate with amiloride + isoproterenol (10 µM). The potential difference will be monitored in actively inflamed areas as judged by endoscopy in comparison to an agar-filled reference butterfly electrode placed in the volar aspect of the forearm. A stable potential with the mean value of a 10-s scoring interval after perfusion of each solution will be recorded by a blinded investigator.

SUMMARY:
The purpose of this study is to establish the novel endoscopically-directed sinus potential difference (EDSPD) assay as an endpoint for therapy of sinus disease.

DETAILED DESCRIPTION:
The purpose of this study is to establish the novel endoscopically-directed sinus potential difference (EDSPD) assay as an endpoint for therapy of sinus disease. This assay provides a means to measure Cl- secretion across the sinus epithelium in human subjects with chronic rhinosinusitis (CRS) and test the relationship between this data and endoscopic findings of inflammation. The technique is appropriate for investigating acquired CFTR dysfunction in sinus epithelium and examining the therapeutic potential of CFTR potentiators for CRS.

ELIGIBILITY:
Patient eligibility criteria are designed to limit enrollment otherwise healthy individuals who are scheduled for standard-of-care nasal endoscopy in the clinic or sinus/skull base surgery.

Inclusion criteria:

* Age > 18 years
* Able to give consent
* A diagnosis of CRS, as determined by the Sinus and Allergy Health Partnership criteria
* Has cultured out at least one gram negative bacteria (e.g. Pseudomonas aeruginosa, Escherichia coli, Stenotrophomonas maltophila) within the previous month
* Is scheduled for either routine endoscopic surgery or has previously undergone endoscopic surgery and presents to clinic for routine endoscopic evaluation

Exclusion criteria:

* Age < 18 years
* Unable to give consent
* Active diagnosis of cancer, autoimmune disease, or any know immunodeficiency
* Women who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be derived from those patients presenting to UAB for endoscopic evaluation of CRS, or who present for standard-of-care sinus or skull base surgery.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Ability to measure CFTR difference using EDSPD testing | 3 Years
  To establish the relationship of EDSPD findings with other validated instruments and markers of CRS disease

CONTACTS AND LOCATIONS:
Overall Officials: Brad Woodworth, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No